CLINICAL TRIAL: NCT05923294
Title: Clinical Comparison of Two Different Graft Harvesting Techniques Applied in Localized Gingival Recessions
Brief Title: Two Different Graft Harvesting Techniques Applied in Localized Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ezgi Gürbüz, Assistant professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0043
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2023-07

CONDITIONS: Gingival Recession, Localized; Sensitivity, Tooth; Attachment Loss, Periodontal
MeSH Terms: conditions — Gingival Recession; Dentin Sensitivity; Periodontal Attachment Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- De-epithelialized gingival unit graft (Experimental): In this split-mouth randomized controlled trial, the coin toss method will determine test and control groups. In both groups, connective tissue graft with a trapezoidal flap design will be applied to the recession area. To obtain the connective tissue graft, the gingival unit graft will be de-epithelialized in the test group.
  Interventions: Procedure: Coronally advanced flap with connective tissue graft
- De-epithelialized free gingival graft (Experimental): In this split-mouth randomized controlled trial, the coin toss method will determine test and control groups. In both groups, connective tissue graft with a trapezoidal flap design will be applied to the recession area. To obtain the connective tissue graft, the traditional free gingival graft will be de-epithelialized in the control group.
  Interventions: Procedure: Coronally advanced flap with connective tissue graft

INTERVENTIONS:
Procedure: Coronally advanced flap with connective tissue graft — In both groups, connective tissue graft with a trapezoidal flap design will be applied to the recession area.

SUMMARY:
The primary purpose of this study is to compare the root coverage rate of the gingival unit-shaped connective tissue graft, obtained by intraoral de-epithelization, with the traditional de-epithelialized free gingival graft in localized recessions of anterior and premolar teeth. In addition, it is aimed to compare the postoperative gingival thickness between the two techniques. The secondary aim is to search the effects of both techniques on periodontal parameters and to evaluate patient-centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists physical status class 1 and 2 patients,healthy patients
2. Nonsmokers
3. Periodontally healthy patients
4. Localized gingival recessions (Miller I, II, and Cairo I recessions with a depth of recession of at least 2 mm) in anterior and premolar teeth

Exclusion Criteria:

1. Medically compromised patients, especially uncontrolled diabetes
2. Pregnancy, lactation, or suspicion of pregnancy,
3. Poor oral hygiene
4. Recessions associated with caries or restoration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Root coverage percentage | Postoperative 6th month
  The comparison of the postoperative recession depth to the initial recession depth
Gingival thickness | Preoperative and postoperative 6th month
  Gingival thickness in the mid-buccal of the recession defect measured with an endodontic spreader and digital recordings

SECONDARY OUTCOMES:
Recession width | Preoperative and postoperative 6th month
  Recession width measured at the cemento-enamel junction
Probing depth | Preoperative and postoperative 6th month
  Probing depth measured at the mid-buccal of the recession defect
Clinical attachment loss | Preoperative and postoperative 6th month
  Clinical attachment loss measured at the mid-buccal of the recession defect
Keratinized gingiva width | Preoperative and postoperative 6th month
  Mid-buccal gingival width measured with a periodontal probe
Vestibular depth | Preoperative and postoperative 6th month
  The distance from the gingival margin to the greatest concavity of the mucosal fold
Pain perception | Postoperative 1st week
  Visual analog scale where higher scores mean a worse outcome and has a minimum value of 0 and a maximum value of 10
Bleeding related to the procedure | Postoperative 1st week
  Bleeding evaluated by a dichotomous index

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kassab MM, Cohen RE. The etiology and prevalence of gingival recession. J Am Dent Assoc. 2003 Feb;134(2):220-5. doi: 10.14219/jada.archive.2003.0137. PMID 12636127
- [Background] Mythri S, Arunkumar SM, Hegde S, Rajesh SK, Munaz M, Ashwin D. Etiology and occurrence of gingival recession - An epidemiological study. J Indian Soc Periodontol. 2015 Nov-Dec;19(6):671-5. doi: 10.4103/0972-124X.156881. PMID 26941519
- [Background] Kassab MM, Badawi H, Dentino AR. Treatment of gingival recession. Dent Clin North Am. 2010 Jan;54(1):129-40. doi: 10.1016/j.cden.2009.08.009. PMID 20103476
- [Background] Cairo F, Pagliaro U, Buti J, Baccini M, Graziani F, Tonelli P, Pagavino G, Tonetti MS. Root coverage procedures improve patient aesthetics. A systematic review and Bayesian network meta-analysis. J Clin Periodontol. 2016 Nov;43(11):965-975. doi: 10.1111/jcpe.12603. Epub 2016 Sep 16. PMID 27454460
- [Background] Zucchelli G, Tavelli L, Barootchi S, Stefanini M, Rasperini G, Valles C, Nart J, Wang HL. The influence of tooth location on the outcomes of multiple adjacent gingival recessions treated with coronally advanced flap: A multicenter re-analysis study. J Periodontol. 2019 Nov;90(11):1244-1251. doi: 10.1002/JPER.18-0732. Epub 2019 Jul 1. PMID 31177536
- [Background] Allen AL. Use of the gingival unit transfer in soft tissue grafting: report of three cases. Int J Periodontics Restorative Dent. 2004 Apr;24(2):165-75. PMID 15119887
- [Background] Kuru B, Yildirim S. Treatment of localized gingival recessions using gingival unit grafts: a randomized controlled clinical trial. J Periodontol. 2013 Jan;84(1):41-50. doi: 10.1902/jop.2012.110685. Epub 2012 Mar 5. PMID 22390550
- [Background] Sriwil M, Fakher MAA, Hasan K, Kasem T, Shwaiki T, Wassouf G. Comparison of Free Gingival Graft and Gingival Unit Graft for Treatment of Gingival Recession: A Randomized Controlled Trial. Int J Periodontics Restorative Dent. 2020 May/Jun;40(3):e103-e110. doi: 10.11607/prd.4180. PMID 32233187